CLINICAL TRIAL: NCT03505112
Title: The Effect of Goal-directed Hemodynamic Therapy on Clinical Outcomes in Patients Undergoing Radical Cystectomy: : A Randomized Controlled Trial
Brief Title: The Effect of Goal-directed Hemodynamic Therapy in Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1712-125-909
Record Dates: First submitted 2018-04-04; First posted 2018-04-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Bladder Cancer; Radical Cystectomy
Keywords: Goal-directed therapy; stroke volume index
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, double-blind, parallel-group, randomized, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed therapy group (Experimental): The patients in goal-directed therapy (GDT) group will be managed according to the goal-directed therapy protocol during the surgery.
  Interventions: Other: Goal-directed therapy
- Control group (No Intervention): The patients in control group will be managed according to standard perioperative care.

INTERVENTIONS:
Other: Goal-directed therapy — The patients in GDT group will receive intravenous crystalloid fluid or vasopressor or inotropic agent according to the goal-directed therapy protocol utilizing FloTrac / EV1000 clinical platform (Edwards Lifesciences, Irvine, CA, USA).
  After induction of anesthesia, the baseline stroke volume index (SVI) is measured and then 200-250 ml of crystalloid is administered over 5-10 minutes. If SVI increase by ≥10%, 200-250 ml of crystalloid is given repeatedly until the increase in SVI <10%. If SVI does not increase by ≥10% and there is no decrease in mean arterial pressure (MAP), revaluate SVI every 10 minutes. Despite an increase in SVI of <10% after fluid challenge, if a decrease in MAP is accompanied by cardiac index (CI) ≤ 2.5 L/min/m2, dobutamine is administered by continuous infusion. If there is a decrease in MAP but no decrease in CI, start low dose norepinephrine continuous infusion.
  Other Names: GDT
  Arms: Goal-directed therapy group

SUMMARY:
Goal-directed therapy (GDT) has been applied to various clinical settings and has been widely researched recently as a method for perioperative management of patients. Radical cystectomy is a complex surgical procedure in which the bladder is removed, followed by urinary diversion. It is an extensive and time-consuming intervention and has high probability of fluid imbalance and bleeding during surgery. We hypothesized that the application of GDT in these patients would improve clinical postoperative outcomes. Therefore, we will attempt to evaluate improvement of postoperative outcomes after applying GDT protocol based on changes in stroke volume index, cardiac index and mean arterial pressure in radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open radical cystectomy
* Patients with American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* Significant hepatic dysfunction, significant renal dysfunction (estimated glomerular filtration rate <60 ml/min)
* Congestive heart failure (New York Heart Association scores ≥3), Left Ventricular Ejection Fraction < 35%
* Arrhythmia
* Coagulopathy (PT INR >1.5)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2021-10-24 (Actual)

PRIMARY OUTCOMES:
A composite of postoperative complications | through the hospitalization period, an average of 2 weeks
  Total incidence of postoperative complications including gastrointestinal complications, complications of infections, wound complications, cardiac events, thromboembolic complications, genitourinary complications, neurological complications based on the Clavien-Dindo classification for radical cystectomy.

SECONDARY OUTCOMES:
The incidence of postoperative gastrointestinal complications | through the hospitalization period, an average of 2 weeks
  Gastrointestinal complications include ileus, constipation, gastric ulcer, anastomic bowel leak according to the Clavien-Dindo classification for radical cystectomy.
The incidence of postoperative complications of infections | through the hospitalization period, an average of 2 weeks
  Complications of infections include urinary tract infection, sepsis, pneumonia, wound infection according to the Clavien-Dindo classification for radical cystectomy.
The incidence of postoperative wound complications | through the hospitalization period, an average of 2 weeks
  Wound Complications mean wound dehiscence diagnosed clinically and requiring resuturing, according to the Clavien-Dindo classification for radical cystectomy.
The incidence of postoperative cardiac events | through the hospitalization period, an average of 2 weeks
  Cardiac events include myocardial infarction, arrhythmia, congestive heart failure, pulmonary edema and transient brain natriuretic peptide increase (serum brain natriuretic peptide values 100-500 pg/ml) according to the Clavien-Dindo classification for radical cystectomy.
The incidence of postoperative thromboembolic complications | through the hospitalization period, an average of 2 weeks
  Thromboembolic complication means pulmonary embolism evidenced by spiral computerized tomography scanning according to the Clavien-Dindo classification for radical cystectomy.
The incidence of postoperative genitourinary complications | through the hospitalization period, an average of 2 weeks
  Genitourinary complications include renal dysfunction, renal failure, urinary leakage according to the Clavien-Dindo classification for radical cystectomy.
The incidence of postoperative neurological complications | through the hospitalization period, an average of 2 weeks
  Neurological complications mean presence of a de novo focal deficit, confusion/delirium according to the Clavien-Dindo classification for radical cystectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, Select, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wuethrich PY, Burkhard FC, Thalmann GN, Stueber F, Studer UE. Restrictive deferred hydration combined with preemptive norepinephrine infusion during radical cystectomy reduces postoperative complications and hospitalization time: a randomized clinical trial. Anesthesiology. 2014 Feb;120(2):365-77. doi: 10.1097/ALN.0b013e3182a44440. PMID 23887199
- [Background] Pearse RM, Harrison DA, MacDonald N, Gillies MA, Blunt M, Ackland G, Grocott MP, Ahern A, Griggs K, Scott R, Hinds C, Rowan K; OPTIMISE Study Group. Effect of a perioperative, cardiac output-guided hemodynamic therapy algorithm on outcomes following major gastrointestinal surgery: a randomized clinical trial and systematic review. JAMA. 2014 Jun 4;311(21):2181-90. doi: 10.1001/jama.2014.5305. PMID 24842135
- [Derived] Yoon HK, Hur M, Kim DH, Ku JH, Kim JT. The effect of goal-directed hemodynamic therapy on clinical outcomes in patients undergoing radical cystectomy: a randomized controlled trial. BMC Anesthesiol. 2023 Oct 9;23(1):339. doi: 10.1186/s12871-023-02285-9. PMID 37814224